CLINICAL TRIAL: NCT05455372
Title: Analysis of Influencing Factors of Oral Helicobacter Pylori Infection and Oral Related Factors on Gastric Helicobacter Pylori Infection and Eradication Therapy Among the Outpatients of A Tertiary Hospital in Xi'an
Brief Title: Influence of Oral Hp Infection and Oral Related Factors on Gastric Hp Infection and Eradication Therapy
Acronym: Hp
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital of Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2022187
Record Dates: First submitted 2022-07-08; First posted 2022-07-13 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori; Oral hygiene; Dental caries; Risk factor; Saliva Test Cassette
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- oral H. pylori negative and gastric H. pylori negative group (No Intervention): These people are tested negative for C13-urea breath test (C13-UBT) and negative for H. pylori Saliva Test Cassette (HPS).
- oral H. pylori positive and gastric H. pylori negative group (No Intervention): These people are tested negative for C13-urea breath test (C13-UBT) and positive for H. pylori Saliva Test Cassette (HPS).
- oral H. pylori negative and gastric H. pylori positive group (Experimental): These patients are tested positive for C13-urea breath test (C13-UBT) and negative for H. pylori Saliva Test Cassette (HPS),they are given PPI quadruple therapy for 14 days. After 4-6 weeks of completing eradication therapy, 13C-UBT will be performed to confirm the results of gastric H. pylori eradication.At the same time, Patients with successful eradication will be instructed to conduct 13C-UBT examination after 1year to confirm whether the recurrence of gastric H. pylori.
  Interventions: Drug: PPI quadruple therapy
- oral H. pylori positive and gastric H. pylori positive group (Experimental): These patients are tested positive for C13-urea breath test (C13-UBT) and positive for H. pylori Saliva Test Cassette (HPS),they are given PPI quadruple therapy for 14 days. After 4-6 weeks of completing eradication therapy, 13C-UBT will be performed to confirm the results of gastric H. pylori eradication, and the oral H. pylori infection will be re-detected by HPS.At the same time, Patients with successful eradication will be instructed to conduct 13C-UBT examination after 1year to confirm whether the recurrence of gastric H. pylori.
  Interventions: Drug: PPI quadruple therapy

INTERVENTIONS:
Drug: PPI quadruple therapy — PPI quadruple therapy refers to ilaprazole 5mg + amoxicillin 1000mg + clarithromycin 500mg + colloidal bismuth tartrate 220mg bid.
  Arms: oral H. pylori negative and gastric H. pylori positive group; oral H. pylori positive and gastric H. pylori positive group

SUMMARY:
Helicobacter pylori (H. pylori) is closely related to the occurrence of gastric cancer and other diseases. The discovery and eradication of H. pylori is of great significance for the prevention and treatment of related diseases. Oral H. pylori may act as a "reservoir" to cause H. pylori to spread between populations and to cause individual gastric H. pylori infection and recurrence.Understanding the oral and gastric H. pylori infection and influencing factors of the population can provide scientific basis for the formulation of local H. pylori infection prevention strategies.Analyzing the influencing factors of H. pylori eradication in the population can improve the local H. pylori eradication rate and reduce the recurrence of H. pylori infection.Therefore, this study intends to analyze the influence of oral H. pylori infection and oral related factors on gastric H. pylori infection and eradication therapy in outpatients of a tertiary hospital in Xi'an.

DETAILED DESCRIPTION:
Taking 300 dyspepsia patients who will undergo C13-urea breath test (C13-UBT) in the outpatient department of gastroenterology of the Second Affiliated Hospital of Xi'an Jiaotong University from July 2022 to March 2024 as the research subjects. A questionnaire survey on factors related to H. pylori infection will be conducted,which include basic information, eating habits, living environment, and oral care habits.From July 2022 to March 2024, Taking 300 patients who will be diagnosed with gastric H. pylori infection in the Gastroenterology Department of the Second Affiliated Hospital of Xi'an Jiaotong University and receive bismuth quadruple H. pylori eradication therapy as the research subjects.The bismuth quadruple regimen is specifically ilaprazole 5mg + amoxicillin 1000mg + clarithromycin 500mg + colloidal bismuth tartrate 220mg bid for 14 days.The research subjects will be also required to complete a questionnaire survey on factors related to the eradication therapy of gastric H. pylori,the contents of the questionnaire include basic information, living habits, side effects of medication, and compliance.All the above populations will be given H. pylori Saliva Test Cassette (HPS) to detect whether H. pylori infection in the oral cavity, and the oral hygiene score (OHI) and the permanent tooth decay missing fill index (DMF) will be also evaluated and recorded.4-6 weeks after the end of treatment, 13C-UBT will be performed to confirm the results of gastric H. pylori eradication, and the oral H. pylori infection will be re-detected by HPS.The patients with successful eradication therapy of gastric H. pylori will be followed up, and the recurrence of gastric H. pylori will be confirmed by 13C-UBT 1 year later.

ELIGIBILITY:
Inclusion Criteria:

The first stage:Study the prevalence and risk factors of oral and gastric H. pylori infection 1. No obstacle to understanding the content of the questionnaire, and can answer the questions accurately, 2. Voluntarily participate in this research and sign the informed consent. The second stage:Study the status and influencing factors of eradication therapy of oral and gastric H. pylori

1. >18 years old,
2. Initial H. pylori eradication therapy,
3. No obstacle to understanding the content of the questionnaire, and can answer the questions accurately,
4. Agree to perform eradication treatment and receive telephone follow-up, and sign the informed consent.

Exclusion Criteria:

The first stage:Study the prevalence and risk factors of oral and gastric H. pylori infection

1. History of taking proton pump inhibitors (PPI), H2 receptor blockers and bismuth agent within two weeks before enrollment,
2. History of taking antibiotics and Chinese medicines with antibacterial effect within one month before enrollment,
3. Complete or partial gastrectomy,
4. Edentulous. The second stage:Study the status and influencing factors of eradication therapy of oral and gastric H. pylori

1. Allergic to penicillin, clarithromycin, ilaprazole, colloidal bismuth tartrate, 2. Complete or partial gastrectomy, 3. Oral scaling within 6 months, 4. Edentulous.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2022-07-08 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Oral and gastric H. pylori infection rate | 1 year
  The gastric infection rate is defined as the proportion of patients diagnosed positive among all subjects undergoing 13-UBT,The oral infection rate is defined as the proportion of patients diagnosed positive among all subjects undergoing HPS.(On the 13-UBT,if the result DOB≥4. 0‰, it can be determined that the subject is gastric H. pylori positive; DOB <4. 0‰,the subject is gastric H. pylori negative.On the HPS,If the T line and C line appear, it is judged to be positive for oral H. pylori infection, but if the C line appears, it is judged to be negative for oral H. pylori infection. If the C line does not appear, it is an invalid test result and needs to be re-tested.)
The affecting factors of oral and gastric H. pylori infection. | 1 year
  Questionnaire used in this study refers to"National Helicobacter pylori Research Questionnaire", which is designed by the Department of Epidemiology and Health Statistics, Peking University School of Medicine.And the questionnaire includes general situation, basic situation, living environment and living habits, personal disease history, related symptoms,and family history, etc.Oral hygiene is assessed using the Simplified Oral Hygiene Index (OHI-S), which is the sum of the Simplified Debris Index (DI-S) and the Simplified Calculus Index (CI-S).Dental caries is measured by the decay missing fill index (DMF),which refers to the sum of caries, lost and filled teeth.Through logistic regression analysis to calculate OR value and P value, to understand the relationship between oral and gastric H. pylori infection and the factors.
Oral and gastric H. pylori eradication rate | 1 year
  The gastric H. pylori positive patients receive PPI quadruple therapy,and after 4-6 weeks of completing eradication therapy, 13C-UBT and HPS are performed.The gastric H. pylori eradication rate is defined as the ratio of the number of subjects who become negative through 13C-UBT after taking the eradication drug to the number of all subjects who take the eradication drug.The oral H. pylori eradication rate is defined as the proportion of subjects taking the eradication drug from positive to negative HPS results.
The affecting factors of gastric H. pylori eradication. | 1 year
  Questionnaire used in this study refers to "National Helicobacter pylori Research Questionnaire", which is designed by the Department of Epidemiology and Health Statistics, Peking University School of Medicine.And the questionnaire includes general situation, basic situation, living environment and living habits, personal disease history, related symptoms, family history,side effects of medication, and compliance etc.Oral hygiene is assessed using the Simplified Oral Hygiene Index (OHI-S), which is the sum of the Simplified Debris Index (DI-S) and the Simplified Calculus Index (CI-S)..Dental caries is measured by the decay missing fill index (DMF),which refers to the sum of caries, lost and filled teeth.Through logistic regression analysis to calculate OR value and P value, to understand the relationship between gastric H. pylori eradication failure and the factors.

CONTACTS AND LOCATIONS:
Overall Officials: Ping Zhao, MD, Principal Investigator — Second Affiliated Hospital of Xi'an Jiaotong University
Locations (1):
- The second affiliated hospital of Xi'an Jiaotong university, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No